CLINICAL TRIAL: NCT01665781
Title: Randomized, Controlled Trial of Erythropoietin in the Prevention of Acute Mountain Sickness
Brief Title: Erythropoietin in the Prevention of Acute Mountain Sickness
Acronym: EPO-AMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ulsan (Other)
Collaborators: HK inno.N Corporation (Industry)
Responsible Party: Principal Investigator, Soon Bae Kim, M.D., PhD., Professor of Medicine, University of Ulsan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMCIRB2012-0534
Record Dates: First submitted 2012-08-12; First posted 2012-08-15 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Acute Mountain Sickness
Keywords: Hemoglobin; Erythropoietin; Acute Mountain sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythropoietin (Experimental): Erythropoietin 10,000U, weekly, for 4 weeks Last dose: 1 week before departure (10days before high altitude)
  Interventions: Drug: Erythropoietin
- Control (No Intervention): No erythropoietin

INTERVENTIONS:
Drug: Erythropoietin
  Arms: Erythropoietin

SUMMARY:
Acute mountain sickness (AMS) is a syndrome of nonspecific symptoms and is therefore subjective. The Lake Louise Consensus Group defined acute mountain sickness as the presence of headache in an unacclimatized person who has recently arrived at an altitude above 2,500 m plus the presence of one or more of the following: gastrointestinal symptoms (anorexia, nausea, or vomiting), insomnia, dizziness, and lassitude or fatigue. An increase in RBC mass is a natural feature of altitude acclimatization. Hypoxia-induced erythropoietin (EPO) secretion begins hours after ascent and stimulates bone marrow production of red blood cells, but this takes weeks to effect an increase in red cell mass . Therefore, it is feasible that EPO therapy weeks before altitude exposure decrease high altitude illness.

In 1996, Young et al in U.S. Army Research Institute of Environmental Medicine (USARIEM) reported that autologous erythrocyte infusion did not ameliorate the decrement in maximal oxygen uptake at 4,300m altitude despite increasing arterial oxygen carrying capacity. On the basis of this report, USARIEM did not recommend use of recombinant EPO for altitude acclimatization.

However, increases in erythrocyte count, hematocrit and hemoglobin associated with EPO therapy have been shown to decrease fatigue and increase work capacity and exercise tolerance. In addition, improvement in CNS function and cognitive ability has been noted with EPO therapy. Subjective benefits include improvement in sleep habits, tolerance to cold; decreased dyspnea, anginal symptoms and tachycardia and improved appetite, all of which are symptoms associated with high altitude illness.

The investigators also reported improved muscle energy metabolism with EPO in dialysis patients, but not with RBC transfusion.

In this study, the investigators will conduct a randomised controlled trial to assess the effect of EPO administration on AMS at an altitude of 4,130 m.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* History of serious illness
* Current smoker or Hemoglobin >15.5gm/dL
* Uncontrolled hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Acute mountain sickness score | At 3230m and 4,130m(Annapurna base camp)
  The AMS self-report score is the sum of answers to five questions (headache; gastrointestinal symptoms (anorexia, nausea, or vomiting); fatigue or weakness; dizziness or lightheadedness; difficulty sleeping) rating from 0 to 3.

SECONDARY OUTCOMES:
Criteria for immediate descent[USARIEM] | At 3230m and 4,130m(Annapurna base camp)
  1. High altitude cerebral edema 1) Mental confusion 2) Ataxia 3) Severe lassitude
  2. Moderate high altitude pulmonary edema 1) Symptoms of dyspnea, weakness, fatigue with mild exertion 2) Cannot perform light activity 3) Headache with cough, dyspnea at rest 4) Heartbeats per min: 110-120 5) Breaths per min: 20-30
  3. Severe AMS: LLS >8

CONTACTS AND LOCATIONS:
Overall Officials: Soon Bae Kim, M.D., Ph.D., Principal Investigator — University of Ulsan
Locations (1):
- Soon Bae Kim, M.D., Ph.D., Seoul, South Korea

REFERENCES:
- [Derived] Heo K, Kang JK, Choi CM, Lee MS, Noh KW, Kim SB. Prophylactic effect of erythropoietin injection to prevent acute mountain sickness: an open-label randomized controlled trial. J Korean Med Sci. 2014 Mar;29(3):416-22. doi: 10.3346/jkms.2014.29.3.416. Epub 2014 Feb 27. PMID 24616593